CLINICAL TRIAL: NCT07186517
Title: Assessment of Key Genetic vaRianTs and thEir iMpacts In Stroke
Brief Title: Genetic Variants in Stroke
Acronym: ÁRTEMIS-Brasil
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Moinhos de Vento (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Other Study IDs: 86795025.0.1001.5330
Record Dates: First submitted 2025-09-09; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Genetic Association Studies
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stroke is the leading cause of death and disability in Brazil and worldwide, with a significant socioeconomic impact. Despite advances in prevention and treatment, the role of genetic variants in ischemic stroke remains underexplored, especially in genetically diverse populations like Brazil's. International studies such as MEGASTROKE and GIGASTROKE have identified risk loci for stroke, but with low representation of the Latin American population. This study aims to fill that gap by evaluating the prevalence and clinical impact of genetic polymorphisms previously described in Brazilians, thereby laying the groundwork for precision medicine within Brazil's Unified Health System (SUS).

DETAILED DESCRIPTION:
Study Overview: ÁRTEMIS-Brazil is a multicenter, case-control study that will recruit 1,000 participants (500 stroke patients and 500 controls) across 10 hospitals in Brazil. All participants will be extensively phenotyped, including demographic, clinical, lifestyle, neuroimaging, and laboratory data, in order to create a comprehensive dataset that links genomic information with health outcomes. Peripheral blood samples will be collected and processed under strict biobanking standards. DNA will undergo whole genome sequencing (WGS), enabling high-resolution investigation of genetic variation in an admixed population.

2) Genomic and Bioinformatics Methodology: The analytical workflow has been designed to ensure high-quality, reproducible results and includes the following components: Pre-processing Removal of adapters, low-quality bases, and contaminant sequences. Filtering of reads based on Phred quality scores to retain only high-confidence sequences.

Alignment and Assembly Mapping of cleaned reads to the human reference genome (GRCh38). Evaluation of coverage, depth, and mapping accuracy. Quality metrics will be benchmarked against international standards.

Variant Analysis Identification and annotation of genetic variants, including single nucleotide polymorphisms (SNPs) and insertions/deletions (indels).

Annotation pipelines (e.g., GATK, ANNOVAR, VEP) will classify variants by predicted functional effect, population frequency, and pathogenicity.

Integration with reference databases such as gnomAD, ClinVar, PharmGKB, and dbSNP to contextualize findings.

Ancestry Analysis Estimation of genetic ancestry proportions using population-specific markers. Adjustment for population stratification in association analyses. Exploration of ancestry contributions to stroke susceptibility and clinical outcomes in Brazil's admixed population.

Pharmacogenetic Analysis Evaluation of variants in genes related to drug metabolism, efficacy, and toxicity (e.g., CYP450 family, platelet receptor pathways, anticoagulant metabolism).

Analysis of implications for treatment of acute ischemic stroke and secondary prevention, with emphasis on tailoring therapy to genetic profiles.

3) Scientific and Clinical Impact: By combining genomic data with detailed phenotypic information, ARTEMIS-Brazil is uniquely positioned to: Identify novel genetic variants associated with stroke in an underrepresented population; Validate known variants in the context of Brazilian admixture; Characterize the contribution of ancestry to stroke risk and outcomes; Generate pharmacogenetic evidence to support personalized stroke care.

The project will advance global understanding of stroke genetics and contribute to the implementation of precision medicine strategies within the Brazilian Unified Health System (SUS). By ensuring representation of admixed populations in genomic research, ÁRTEMIS-Brazil will fill a major gap in current knowledge and create a foundation for more equitable healthcare.

ELIGIBILITY:
Inclusion Criteria:

Cases

* Age ≥18 years;
* Confirmed diagnosis by neuroimaging (CT or MRI) of a first episode of ischemic stroke in the last 12 months;
* TOAST classification of stroke available: cardioembolic, lacunar, atherosclerotic, or undetermined due to the presence of multiple sources (cardioembolic/atherosclerotic);
* Modified Rankin Scale (mRS) ≤4 at the time of inclusion;
* Ability and willingness to provide consent and participate in follow-up assessments.

Controls

* Age ≥18 years;
* Reside in the same household or, if not, in the same neighborhood as the case group participant;
* Not be a blood relative of the case group participant;
* Ability and willingness to provide consent and participate in follow-up assessments.

Exclusion Criteria:

Cases

* Ischemic stroke with a distinct etiology based on TOAST criteria (e.g., infectious, autoimmune, endocarditis, reversible cerebral vasoconstriction syndrome, drug-related causes);
* Diagnosis of monogenic or mitochondrial disorders, such as CADASIL, Fabry disease, homocystinuria, MELAS, sickle cell disease, among others;
* Clinical conditions that reduce life expectancy to less than one year (e.g., neoplasia);
* Inability to undergo magnetic resonance imaging (due to metal artifacts, MRI-incompatible implants, claustrophobia);
* Other conditions that, at the investigator's discretion, prevent participation or compromise follow-up.

Controls

* Personal history of stroke, transient ischemic attack (TIA), coronary, or peripheral artery disease;
* Serious comorbidities that may impact participation or confound the results;
* Clinical conditions that reduce life expectancy to less than one year;
* Inability to provide consent due to cognitive impairment or other factors;
* Inability to undergo magnetic resonance imaging (due to metal artifacts, incompatible implants, claustrophobia);
* Diagnosis of monogenic or mitochondrial disorders, such as CADASIL, Fabry disease, homocystinuria, MELAS, or sickle cell disease;
* Other conditions that, at the investigator's discretion, prevent participation or compromise follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 500 ischemic stroke patients and 500 controls with no family or personal history of stroke.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of stroke-related genetic polymorphisms measured by whole genome sequencing (WGS) | 60 months
  Frequency and distribution of single nucleotide polymorphisms (SNPs) and small insertions/deletions (indels) previously associated with stroke, identified from whole genome sequencing data. Frequencies will be compared with international genomic databases to evaluate similarities and differences in an admixed Brazilian population. Unit of Measure: Percentage of participants carrying the variant; allele frequency (%).
Genetic ancestry composition assessed by whole genome sequencing (WGS) | 60 months
  Proportion of ancestry components (e.g., European, African, Indigenous American) estimated from population-specific genetic markers using WGS. Comparison between stroke cases and controls will be performed to explore associations with stroke risk. Unit of Measure: Proportion of ancestry components (%).
Pharmacogenetic variants associated with drug metabolism identified by whole genome sequencing (WGS) | 60 months
  Prevalence of variants in pharmacogenes (e.g., CYP450 genes, platelet receptor genes, anticoagulant metabolism pathways) assessed through WGS. Results will be compared with reference databases and analyzed in stroke cases and controls. Unit of Measure: Percentage of participants carrying pharmacogenetically relevant variants; allele frequency (%).

CONTACTS AND LOCATIONS:
Overall Officials: Ana C de Souza, PhD, Principal Investigator — Hospital Moinhos de Vento
Locations (11):
- Brazil (11):
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ophir Loyola, Belém
  - Hospital Metropolitano Dr. Célio de Castro, Belo Horizonte
  - Hospital Geral de Roraima, Boa Vista
  - Hospital Universitário Maria Aparecida Pedrossian, Campo Grande
  - Hospital Geral de Fortaleza, Fortaleza
  - Clínica Neurológica, Joinville
  - Hospital Geral de Palmas, Palmas
  - Hospital da Restauração Governador Paulo Guerra, Recife
  - Hospital Universitário Edgar Santos, Salvador
  - Hospital São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided